CLINICAL TRIAL: NCT06340607
Title: Impact of Neohepatic Albumin-Bilirubin Scores on Renal Outcomes Following Living-donor Liver Transplantation: Propensity Score Analysis
Brief Title: Neohepatic Albumin-Bilirubin Scores on Renal Outcomes in Living-donor Liver Transplantation Recipients
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Jun-Gol Song, Professor, Asan Medical Center
Other Study IDs: 2023-0561
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Acute Kidney Injury; Chronic Kidney Diseases; Graft Failure
MeSH Terms: conditions — Acute Kidney Injury; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Recipients with neohepatic ALBI ≥ -1.615: The ALBI score was calculated using the formula: (log10bilirubin × 0.66) + (albumin × -0.085), where bilirubin is measured in μmol/L and albumin in g/L. Recipients with neohepatic (post-reperfusion) ALBI ≥ -1.615
- Recipients with neohepatic ALBI < -1.615: Recipients with neohepatic (post-reperfusion) ALBI < -1.615

SUMMARY:
This study investigates the association between post-reperfusion (neohepatic) ALBI scores and post-LT renal outcomes in living-donor LT (LDLT) recipients.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) after liver transplantation (LT) significantly affects patient and graft outcomes. The Albumin-Bilirubin (ALBI) score, an objective and sensitive index of liver function, has potential applicability in predicting outcomes following LT. This study investigates the association between post-reperfusion (neohepatic) ALBI scores and post-LT renal outcomes in living-donor LT (LDLT) recipients.

ELIGIBILITY:
Inclusion Criteria:

* living donor liver transplantation recipients (≥18 years)

Exclusion Criteria:

* preoperative serum creatinine (sCr) > 1.4 mg/dL, diagnosed CKD or hepatorenal syndrome (HRS), or hemodialysis at baseline

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: living donor liver transplantation recipients at Asan Medical Center, Seoul, Korea from January 2012 to December 2019
Sampling Method: Non-Probability Sample
Enrollment: 3422 (Actual)
Dates: Start 2012-01-05 (Actual); Primary Completion 2020-01-05 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
acute kidney injury | within 7 days after surgery
  determined by change in sCr according to the Kidney Disease: Improving Global Outcomes (KDIGO) definition (increase in sCr of ≥26.5 mmol litre-1 within 48h or ≥1.5 times baseline within 7 days after surgery

SECONDARY OUTCOMES:
chronic kidney injury | within 1 year after surgery
  when renal function assessed by calculating estimated serum glomerular filtration using the abbreviated modification of diet in renal disease equation was <60 mL/min/1.73 m2 for 3 months or more, irrespective of cause
graft failure | the graft failure at overall period (calculated from the date of surgery to the last follow-up) from the date of surgery (up to 10 years)]
  graft failure

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, Song-pa Gu, South Korea

IPD SHARING:
Plan to Share IPD: No